CLINICAL TRIAL: NCT04767776
Title: Non Inferiority Study of a Reduced Dose of Activated Charcoal on Rivaroxaban Pharmacokinetics.
Acronym: RICHAR2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 18CH050; 2019-004425-25 (EudraCT Number)
Record Dates: First submitted 2021-02-19; First posted 2021-02-23 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Healthy
Keywords: Rivaroxaban,; Activated charcoal; Pharmacokinetics; Poisoning
MeSH Terms: conditions — Anthrax; Poisoning | interventions — Rivaroxaban; Charcoal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A (Experimental): * Period " rivaroxaban and 6 milligram of activated charcoal "
  * Washout period (6 days)
  * Period " rivaroxaban and 12 milligram of activated charcoal "
  * Washout period (6 days)
  * Period " rivaroxaban and 50 milligram of activated charcoal "
  * Washout period (6 days)
  Interventions: Drug: Rivaroxaban; Drug: Activated charcoal
- Arm B (Experimental): * Period " rivaroxaban and 12 milligram of activated charcoal "
  * Washout period (6 days)
  * Period " rivaroxaban and 6 milligram of activated charcoal "
  * Washout period (6 days)
  * Period " rivaroxaban and 24 milligram of activated charcoal "
  * Washout period (6 days)
  Interventions: Drug: Rivaroxaban; Drug: Activated charcoal
- Arm C (Experimental): * Period " rivaroxaban and 50 milligram of activated charcoal "
  * Washout period (6 days)
  * Period " rivaroxaban and 24 milligram of activated charcoal "
  * Washout period (6 days)
  * Period " rivaroxaban and 6 milligram of activated charcoal "
  * Washout period (6 days)
  Interventions: Drug: Rivaroxaban; Drug: Activated charcoal
- Arm D (Experimental): * Period " rivaroxaban and 24 milligram of activated charcoal "
  * Washout period (6 days)
  * Period " rivaroxaban and 50 milligram of activated charcoal "
  * Washout period (6 days)
  * Period " rivaroxaban and 12 milligram of activated charcoal "
  * Washout period (6 days)
  Interventions: Drug: Rivaroxaban; Drug: Activated charcoal

INTERVENTIONS:
Drug: Rivaroxaban — rivaroxaban 40 mg/day (1 day).
Drug: Activated charcoal — Activated charcoal 2 hours after rivaroxaban administration (1 day).

SUMMARY:
Rivaroxaban is a direct oral anticoagulant that target specifically activated factor X. Bleeding events related to rivaroxaban are the consequence of physiopathologic, pharmacokinetic issues or poisoning. A recent study, in healthy subjects, shows that activated charcoal can reduce significantly exposition to rivaroxaban. However, no results are available on the minimal dose of activated charcoal necessary in rivaroxaban poisoning. The objective of this study is to evaluate the effect of 4 dosing regimen activated charcoal on rivaroxaban pharmacokinetics. It corresponds to a randomised open trial with an incomplete cross over design (3 occasions). It will enrol 12 healthy subjects. Four treatments modalities will be studied: rivaroxaban with 50g, 24g, 12g and 6g of activated charcoal administrated 3 hours after rivaroxaban intake.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated or beneficiary of a social security category
* Having signed the inform consent form
* Having signed the biologic consent form
* Men aged between 18 and 40 years
* Weight between 55 and 92 kilogram
* normal clinical exam
* normal biological exam

Exclusion Criteria:

* Contra-indication to rivaroxaban
* Contra-indication to activated charcoal
* With a history of hemorrhagic disease
* Smoker
* Organic lesion likely to bleed
* Severe liver disease
* Severe kidney failure
* Gastroduodenal ulcers
* Any medication taken during the week prior to the start of the study
* Consumption of grapefruit juice
* Routine ingestion of excessive amounts of coffee, tea, chocolate and/or caffeinated beverages
* Practice of violent sports
* Fructose intolerance
* Glucose-galactose malabsorption syndrome or sucrase-isomaltase deficiency syndrome
* Notable medical history (cardiovascular pathology, pulmonary, neurology ...)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
plasma concentrations of rivaroxaban | 1, 2, 2.5, 3, 3.5, 4, 5, 7, 9, 12, 24 hours after rivaroxaban administration
  rivaroxaban pharmacokinetics

SECONDARY OUTCOMES:
Adverse events | 24 hour after rivaroxaban administration
  Analysis adverse events related to the administration of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick MISMETTI, MD PhD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No